CLINICAL TRIAL: NCT01196884
Title: IMMUNE-GENETIC ASSESSMENT OF PRIMARY ITP IN ADULT
Brief Title: Immune Thrombocytopenia (ITP) Immune-Genetic Assessment
Acronym: UNIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Sanitaria-Universitaria Integrata di Udine (Other)
Responsible Party: Francesco Zaja, Clinica Ematologica, Azienda Ospedaliero Universitaria S. Maria Misericordia di Udine
Other Study IDs: UNIT
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2010-09

CONDITIONS: Thrombocytopenia
Keywords: Patients with primary Immune Thrombocytopenia (ITP)
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Asymptomatic ITP patients
- ITP patients treated with Rituximab
- ITP patients treated with steroids

SUMMARY:
Primary ITP has wide heterogenous biology, presentation and response to therapy.

The immune-genetic assessment of ITP may help to identify differences among patients with ITP and optimize the therapeutic choice.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with primary ITP

Exclusion Criteria:

* Secondary ITP

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2010-09

CONTACTS AND LOCATIONS:
Locations (13):
- Italy (13):
  - Istituto di Ematologia L. & A. Seragnoli, Bologna
  - Department of Hematology and Bone Marrow Transplantation Unit, Oncology Center Armando Businco, Cagliari
  - UF Ematologia, Policlinico di Careggi, Florence
  - U.O. Ematologia 2, IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - Department of Oncology/Haematology, Niguarda Ca'Granda Hospital, Milan
  - Clinica Ematologica, Dipartimento di Medicina Clinica e Sperimentale, Università degli Studi del Piemonte Orientale "Amedeo Avogadro, Novara
  - Istituto di Immunologia, Dipartimento di Scienze Mediche dell'Università degli Studi del Piemonte Orientale "Amedeo Avogadro", Novara
  - Department of Medical and Surgical Sciences, University of Padova, Padua
  - Oncology-Hematology Department, "S. Maria delle Croci" Hospital, Ravenna
  - Institute of Hematology, Catholic University,, Roma
  - Ematologia, Ospedale Ca' Foncello, Treviso
  - Clinica Ematologica AOUD S. Maria Misericordia, Udine
  - Ematologia, San Bortolo Hospital, Vicenza